CLINICAL TRIAL: NCT05231382
Title: A Prospective, Multicenter, Phase III Clinical Study Comparing Continuous Hepatic Arterial Infusion of Raltetrexed With Oxaliplatin(SALOX) Versus FOLFOX in Advanced Hepatocellular Carcinoma
Brief Title: Hepatic Arterial Infusion of Raltetrexed With Oxaliplatin(SALOX) Versus FOLFOX in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Associate Director of Minimally Invasive Intervention, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-380-01
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: SALOX; Arterial infusion chemotherapy; FOLFOX; Raltetrexed; Oxaliplatin; Fluorouracil; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — raltitrexed; Oxaliplatin; Therapeutics; Fluorouracil; Leucovorin; Folfox protocol

STUDY DESIGN:
Intervention Model Description: Oxaliplatin retitrexed
Masking Description: Oxaliplatin Fluorouracil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group SALOX regimen (Experimental): The therapeutic scheme was SLAOX regimens including oxaliplatin (130 mg/m2 infusion for 3 hours on day 1), Raltitrexed (2mg/m2 infusion for 30-60 minutes on day 1)
  Interventions: Procedure: Raltitrexed, oxaliplatin (SALOX) treatment
- Control group FOLFOX regimen (Active Comparator): The therapeutic scheme was modified FOLFOX6 regimens including oxaliplatin (130 mg/m2 infusion for 3 hours on day 1), leucovorin (200 mg/m2 from hour 3 to 5 on day 1) and Fluorouracil (400 mg/m2 in bolus, and then 2,400 mg/m2 continuous infusion 46 hours).
  Interventions: Procedure: Oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment

INTERVENTIONS:
Procedure: Raltitrexed, oxaliplatin (SALOX) treatment — Hepatic arterial infusion (HAI) of Raltitrexed, oxaliplatin (SALOX) treatment
  Arms: Experimental group SALOX regimen
Procedure: Oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment — Hepatic arterial infusion (HAI) of oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment
  Arms: Control group FOLFOX regimen

SUMMARY:
Hepatic artery infusion chemotherapy (HAIC) have shown promising outcomes in patients with advanced hepatocellular carcinoma (HCC).In China, Oxaliplatin combined with 5-fluorouracil is commonly used in continuous hepatic arterial perfusion chemotherapy.But the 5-FU requiring a long infusion and Calcium folate is also needed to sensitize 5-FU. Moreover, 5-FU regimen was associated with a variety of adverse events, which limited its application in HAIC.Compared to 5-fluorouracil, raltetrexed is less toxic, has a stronger anti-tumor effect and can be administered in just two to three hours. However, the comparison of the two drugs in HAIC to treat advanced HCC has not been reported. In this study, we will evaluate the the progression-free survival(PFS)、objective response rate（ORR）、 disease vacancy rate（DCR）、overall survival (OS) and safety in patients with advanced hepatocellular carcinoma (Ad-HCC) who are undergoing hepatic arterial infusion (HAI) of Raltetrexed plus oxaliplatin (SALOX) compared with oxaliplatin, fluorouracil/leucovorin (FOLFOX) treatment by designing prospective, multi-center phase III clinical study.

DETAILED DESCRIPTION:
Femoral artery puncture and catheterization were performed in every cycle of treatment,a micro-catheter was inserted and located in feeding hepatic artery. The therapeutic scheme was that, the experimental group SALOX regimen including oxaliplatin (130 mg/m2 infusion for 3 hours on day 1) and raltetrexed (2mg/m2 for 30 to 60 minutes on day 1) . The control group modified FOLFOX6 regimens including oxaliplatin (130 mg/m2 infusion for 3 hours on day 1), leucovorin (200 mg/m2 from hour 3 to 5 on day 1) and Fluorouracil (400 mg/m2 in bolus, and then 2,400 mg/m2 continuous infusion 46 hours). All chemo-drugs were given by HAI. Treatment was repeated every 3 weeks and continued until intrahepatic lesions progression or unacceptable toxicity.Enhanced CT or MRI was performed every 6 weeks after treatment begins. Routine follow-up intervals were 2-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form (ICF) and any locally required authorization obtained from the patient prior to any mandatory study specific procedures, sampling, and analyses.
* Provision of signed and dated written genetic informed consent prior to optional collection of sample for genetic analysis.
* Patients with BCLC stage C hepatocellular carcinoma confirmed by pathology or clinically diagnosed
* Age ≥18 years and < 75 years at the time of screening.
* Portal vein invasion or extrahepatic oligosaccharides were detected by baseline imaging. Oligosaccharides were defined as no more than two extrahepatic organs and no more than three tumors.
* Child-Pugh score class A to B
* No local antitumor therapy for hepatocellular carcinoma was received within 4 weeks prior to enrollment
* No previous systemic antitumor therapy for hepatocellular carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* The expected survival time is no less than 3 months
* Patients with HBV infection, which is characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥10 IU/ml or above the limit of detection per local lab standard), must be treated with antiviral therapy, as per institutional practice. HBV antiviral therapy must be initiated prior to randomization and patients must remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication. Patients must show evidence HBV stabilization or signs of viral response (e.g., reduction HBV DNA levels) prior to starting IP. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/ml or under the limit of detection per local lab standard) do not require anti-viral therapy prior to randomization. These subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥10 IU/ml or above the limit of detection per local lab standard). HBV DNA detectable subjects must initiate and remain on antiviral therapy for the study duration and for 6 months after the last dose of study medication.
* Patients with HCV infection must have management of this disease per local institutional practice throughout the study. HCV diagnosis is characterized by the presence of detectable HCV ribonucleic acid (RNA) or anti-HCV antibody upon enrollment.
* At least 1 measurable intrahepatic lesion suitable for repeat assessments according to the following mRECIST criteria: （1）Liver lesions that show typical features of HCC on IV contrast-enhanced CT or MRI scans, ie, hypervascularity in the arterial phase with washout in the portal or the late venous phase；（2）Viable, non-necrotic portion (arterial phase IV contrast-enhancing) that can be accurately measured at baseline as ≥10 mm in the longest diameter.
* Adequate organ and marrow function as defined below. Criteria "a," "b," "c," and "f" may not be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

Hemoglobin ≥9.0 g/dL、Absolute neutrophil count ≥1000/µL、Platelet count ≥50000/µL、Total bilirubin ≤2.0 × the upper limit of normal (ULN)、alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 × ULN、Albumin ≥2.8 g/dL、International normalized ratio ≤1.6、2+ proteinuria or less urine dipstick reading、Calculated creatinine clearance (CL) ≥30 mL/min as determined by Cockcroft-Gault (using actual body weight) or 24hour urine creatinine CL

Males:

Creatinine CL = Weight (kg) × (140 - Age) (mL/min) 72 × serum creatinine (mg/dL)

Females:

Creatinine CL = Weight (kg) × (140 - Age) × 0.85 (mL/min) 72 × serum creatinine (mg/dL)

* Must have a life expectancy of at least 12 weeks.
* Body weight >30 kg

Exclusion Criteria:

* A history of liver decompensation, such as refractory ascites, gastrointestinal bleeding, or hepatic encephalopathy; Uncontrolled complications, including but not limited to: Persistent or activity (except the HBV and HCV) infection, symptoms of congestive heart failure and uncontrolled diabetes, uncontrolled hypertension, unstable angina, uncontrolled arrhythmias, active ILD, severe chronic GI disease accompanied by diarrhea, or compliance with requirements may limit the research, resulted in significant increase risk of AE or influence Subjects provided psychiatric/social problem status on their ability to provide written informed consent.A history of active primary immunodeficiency or human immunodeficiency virus; Active or previous records of autoimmune disease or inflammatory diseases, including inflammatory bowel disease (e.g., colitis or crohn's disease], diverticulitis, except [diverticulosis], systemic lupus erythematosus (sle), sarcoidosis syndrome or wegener syndrome (e.g., granulomatous vasculitis, gray's disease, rheumatoid arthritis, the pituitary gland inflammation and uveitis]).
* Known to produce allergic or hypersensitive reactions to any study drug or any excipient thereof;
* Significant clinical gastrointestinal bleeding or a potential risk of bleeding was identified by the investigator during the 30 days prior to study entry.
* Tumors of the central nervous system, including metastatic brain tumors;
* Pregnant women or breast-feeding patients;
* Complicated with other malignant tumors:

  * Malignant tumors that have been treated for therapeutic purposes, have no known active disease for ≥5 years prior to the first administration of the study drug, and have a low potential risk of recurrence
  * Fully treated non-melanoma skin cancer or malignant freckle moles with no evidence of disease
  * Fully treated carcinoma in situ without evidence of disease
* Prior to the initial dosing of the study drug, they had received anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy
* HAIC treatment was received prior to initial dosing of the study drug
* Has received anti-tumor system therapy for HCC. Non-anti-tumor purpose combined hormone therapy (e.g., hormone replacement therapy) is excluded.
* Is currently using, or has used an immunosuppressive drug within 14 days prior to the first dose of the investigational drug. This standard has the following exceptions:

  * intranasal, inhaled, topical or topical steroids (e.g., intraarticular)
  * Systemic corticosteroid therapy not exceeding 10 mg/ day of prednisone or its physiological equivalent as a prophylactic use of steroids for hypersensitivity (e.g., CT scan pretherapy medication)
  * Steroids as a prophylactic for allergic reactions.
* A live attenuated vaccine was administered within 30 days prior to the first administration of the study drug. Note: If enrolled, patients shall not receive live attenuated vaccine within 30 days of receiving study drug therapy and after the last administration of study drug.
* Pregnant or lactating women, or fertile men or women who do not want to use high-efficiency contraceptives, 6 months after the last dosing of study treatment, from screening to study treatment. Based on the patient's preferred and customary lifestyle, abstinence during treatment and washout is an acceptable contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Two-years progression-free survival rate | Two years
  It is defined as the percentage of patients who achieve a time interval of two years of no disease progression (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (by any cause) from date of enrollment, whichever occurs first.

SECONDARY OUTCOMES:
Two-years Overall Survival Rate | Two years
  Percentage of patients who survived two years after inclusion
Objective response rate | Two years
  The percentage of patients who achieved a complete or partial response at some point in their life
Evaluate the patient's cancer-related QoL using the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ), the EORTC QLQ-HCC18. | From date of randomization up to two years, approximately
  Change in sub-scale and total scores of EORTC QLQ-HCC18 from baseline through follow-up.
Evaluate the patient's cancer-related QoL using the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ), the EORTC QLQ-C30. | From date of randomization up to two years, approximately
  Change in sub-scale and total scores of EORTC QLQ-C30 from baseline through follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D. & Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] Lyu N, Lin Y, Kong Y, Zhang Z, Liu L, Zheng L, Mu L, Wang J, Li X, Pan T, Xie Q, Liu Y, Lin A, Wu P, Zhao M. FOXAI: a phase II trial evaluating the efficacy and safety of hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin for advanced hepatocellular carcinoma. Gut. 2018 Feb;67(2):395-396. doi: 10.1136/gutjnl-2017-314138. Epub 2017 Jun 7. No abstract available. PMID 28592441